CLINICAL TRIAL: NCT03795415
Title: Evaluation of the Short- and Mid-term Effects of an Empowerment Program Focused on Serostatus Disclosure Management for Women Living With HIV in Mali
Brief Title: ANRS12373 GUNDO SO - Evaluation of an Empowerment Program for WLHIV in Mali
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Fondation de France (Other); Aix Marseille Université (Other); Université du Québec a Montréal (Other); Centre Population et Développement (CEPED), Paris, France (Unknown); ARCAD-SIDA MALI (Other); Groupe de Recherche en Psychologie Sociale (GRePS), Bron, France (Unknown); Coalition Plus, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: ANRS12373
Record Dates: First submitted 2018-06-15; First posted 2019-01-07 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: HIV Seropositivity; Disclosure; Empowerment; HIV/AIDS
Keywords: WLHIV; empowerment; disclosure; Mali
MeSH Terms: conditions — HIV Seropositivity; Empowerment; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immediate Arm (G1): 3 months after enrollment, each big groups of 16 will be split in two groups. Women in G1 will receive the intervention Gundo-So immediately. (From month 3 to month 6).
  112 women will be in immediate arm in 14 groups of 8 women.
  Interventions: Behavioral: Gundo So
- Delayed Arm (G2): 3 months after enrollment, each big groups of 16 will be split in two groups. Women in G2 will receive the intervention Gundo-So 3 months after. (From month 6 to month 9).
  112 women will be in delayed arm in 14 groups of 8 women.
  Interventions: Behavioral: Gundo So

INTERVENTIONS:
Behavioral: Gundo So — Gundo-So was adapted from a program established in quebec. It has been implemented in Mali following 3 phases: 1) cultural adaptation; 2) validation using a pre-post intervention evaluation; 3) scale-up
  The programm consists on 9 group meetings group spread over 9 weeks (for 8 WLHIV + 2 trained community-based leaders). Each meeting has some particular thematics with adapted tools.
  Other Names: Gundo So - The room of confidences

SUMMARY:
The objective of this research is to measure the short- and mid-term effects of an empowerment program focused on serostatus disclosure management for women living with HIV (WLHIV) in Mali on the "burden of secrecy".

DETAILED DESCRIPTION:
Serostatus disclosure is a critical issue for persons living with HIV (PLHIV). Studies identified numerous benefits associated with disclosure, but various negative consequences have also been documented. Gender inequality must be taken into account regarding the disclosure issue, in particular in Mali, where women are economically dependent and have a low decision-making power. Moreover, in Mali, since 2006, PLHIV have a legal obligation to disclose their serostatus to their spouse and sexual partner(s) " as soon as possible, or within 6 weeks " after the diagnosis. Although this law is not enforced, it highlights the sensitive nature of the serostatus disclosure issue and raise concerns among PLHIV and other stakeholders.

To support women living with HIV (WLHIV), an empowerment program (Gundo-So) was implemented by ARCAD-SIDA in Mali, in collaboration with several partners. This program aims to empower WLHIV, so that they can make informed decision about disclosing or keeping their serostatus secret in their various life contexts, and that they can identify strategies to disclose or to keep the secret, as well as to manage potential negative reactions. Gundo-So ("The room of confidences") was adapted from a program established in quebec and has been implemented in Mali.

The objective of this research is to measure the short- and mid-term effects of an empowerment program focused on serostatus disclosure management for women living with HIV (WLHIV) in Mali on the "burden of secrecy".

The evaluation of the effects of the Gundo-So program will be helpful to assess the relevance of a national or subregional extension of the program, or even an adaptation to other target populations (e.g. heterosexual men and men who have sex with men living with HIV).

ELIGIBILITY:
Inclusion Criteria:

* women living with HIV
* living in Bamako area (Mali)
* over 18 years old
* knowing their serological status for more than 6 months and less than 5 years
* being available to participate in the 9 weekly sessions lasting about 2 hours each.

Exclusion Criteria:

* having already participated in Gundo-So

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The programm Gundo So has been adapted for groups of malian women living with HIV (WLHIV). The study population is described with the inclusion criteria. Moreover, in order to participate at this research, women have to answer "Yes" at at least one of those 2 questions :
  * (1) is it difficult for you to share your HIV serostatus ; and (1.1) is it inconvenient for you?
  * (2) is it difficult for you to keep your HIV serostatus secret; and (2.1) is it inconvenient for you?
Sampling Method: Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Short term evaluation of the burden associated with the disclosure issue using questionnaires | The short term effect will be measured at the end of the intervention and compared between Group 1 and 2. Up to 6 months from the beginning of the randomization to the end of the intervention
  Improvement of the management of the sharing of the serological status. Empowerment in sharing the HIV status (questionnaire)
Short term evaluation of the burden associated with the secrecy issue using questionnaires | The short term effect will be measured at the end of the intervention and compared between Group 1 and 2. Up to 6 months from the beginning of the randomization to the end of the intervention
  Improvement of the management of the secret of the serological status. Empowerment in keeping secret the HIV status (questionnaire)
Mid term evaluation of the burden associated with the disclosure issue using questionnaires | The mid term effect will be measured 9 months after the intervention : up to 9 months after the intervention
  Improvement of the management of the sharing of the serological status. Empowerment in sharing the HIV status (questionnaire)
Mid term evaluation of the burden associated with the secrecy issue using questionnaires | The mid term effect will be measured 9 months after the intervention : up to 9 months after the intervention
  Improvement of the management of the secret of the serological status. Empowerment in keeping secret the HIV status (questionnaire)

SECONDARY OUTCOMES:
Changes in quality of life of WLHIV: questionnaire | Measured at the randomization and then immediately after the intervention
  Assess the changes in quality of life (questionnaire)
Evolution of sexual practices and use of risk reduction strategies | Measured at the randomization and then immediately after the intervention
  Assess changes of sexual practices and risk reductions strategies (questionnaire)
Reported compliance (questionnaire) | Measured at the randomization and then immediately after the intervention
  Assess changes of reported compliance throught HIV antiretroviral treatments (questionnaire)
Biological data : HIV viral load | From 6 months before the intervention until the last follow up (total 2 years)
  Access changes in HIV viral load due to the intervention (via the medical file)
Biological data : cluster of differentiation 4 levels | From 6 months before the intervention until the last follow up (total 2 years)
  Access changes in cluster of differentiation 4 levels due to the intervention (via the medical file)
Satisfaction of the intervention: questionnaire | Measured immediately after the intervention
  Assess the satisfaction of the intervention using questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marie Préau, Pr, Principal Investigator — GRePS
Locations (6):
- Mali (6):
  - CESAC de BAMAKO, Bamako
  - Usac Cnam, Bamako
  - USAC commune IV, Bamako
  - USAC commune I, Bamako
  - USAC commune VI, Bamako
  - USAC commune V, Bamako

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bernier A, Yattassaye A, Beaulieu-Prevost D, Otis J, Henry E, Flores-Aranda J, Massie L, Preau M, Keita BD. Empowering Malian women living with HIV regarding serostatus disclosure management: Short-term effects of a community-based intervention. Patient Educ Couns. 2018 Feb;101(2):248-255. doi: 10.1016/j.pec.2017.07.030. Epub 2017 Jul 26. PMID 28789863